CLINICAL TRIAL: NCT03589846
Title: The Effect of Palatoglossus and Genioglossus Stimulation During Drug-Induced Sleep Endoscopy
Brief Title: Muscle Stimulation During DISE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Kent, Assistant Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 181078
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All patients who meet eligiblity will undergo muscle stimulation at the same time as the operative DISE procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Muscle stimulation (Experimental): Consented participants who meet eligibility will have a drug induced sleep endoscopy (DISE) and the Grass S88 muscle stimulator.
  Interventions: Device: Grass S88 Muscle Stimulator

INTERVENTIONS:
Device: Grass S88 Muscle Stimulator — The Grass S88 nerve and muscle stimulator is a widely-used tool in electromyography and nerve conduction studies. Under anesthesia, fine-wire electrodes will be placed into the right genioglossus muscle (in the floor of the mouth) and the right palatoglossus muscle (in the anterior tonsillar pillar).

SUMMARY:
Drug-induced sleep endoscopy (DISE) is a widely used tool for assessing collapse patterns of the upper airway anatomy during sleep. Hypoglossal nerve stimulation therapy for obstructive sleep apnea suffers from variable response at the level of the soft palate. We propose a study examining the physiologic effect of palatoglossus and genioglossus muscle stimulation during DISE.

DETAILED DESCRIPTION:
This is a single-arm study involving the use of a diagnostic device (muscle stimulator) that is not currently utilized in any clinical decision-making processes for OSA patients. All patients scheduled for DISE as part of their regular clinical care will be screened for enrollment via the previously described inclusion and exclusion criteria. The study is not blinded. No diagnostic information collected from muscle stimulation will be used in clinical decision-making processes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (≥18 years old)
2. A diagnosis of obstructive sleep apnea as determined by polysomnogram with an apnea-hypopnea index of ≥ 5.0/hr.
3. Intolerant of CPAP therapy due to physical or psychosocial limitations as determined by clinical history
4. Scheduled to undergo DISE as part of routine clinical assessment for further evaluation of pharyngeal anatomy

Exclusion Criteria:

1. Unable to consent for research due to a pre-existing neurologic condition as determined by PI
2. Unable to consent for research due to language barriers
3. A history of egg allergy as determined by history or self-reports
4. Currently pregnant as determined by patient report or pre-operative anesthesia evaluation
5. Cardiopulmonary or other medical conditions precluding safe propofol sedation as determined by pre-operative anesthesia evaluation
6. History of palatal or pharyngeal airway surgery including tonsillectomy as determined by clinical history and exam
7. History of radiation treatment to the head or neck as determined by history and/or physical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Basic physiologic measurements | Collected during operative procedure, taking about 15 minutes.
  This study involves the collection of basic physiologic measurements (airway cross-sectional diameter with and without muscle stimulation) during a single session of DISE.

SECONDARY OUTCOMES:
Amount of current needed for adequate stimulation | Collected during operative procedure, taking about 15 minutes.
  Obtain preliminary data regarding including the amount of current needed to adequately stimulate the palatoglossus muscle.

CONTACTS AND LOCATIONS:
Overall Officials: David T. Kent, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashvile, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No